CLINICAL TRIAL: NCT04063631
Title: Pulmonary Epithelial Barrier and Immunological Functions at Birth and in Early Life - Key Determinants of the Development of Asthma
Brief Title: Pulmonary Epithelium, Immunology and Development of Asthma: Breathing Together
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Imperial College London (Other)
Collaborators: Queen Mary University of London (Other); University of Bristol (Other); University of Southampton (Other); University of Edinburgh (Other); Queen's University, Belfast (Other); University of Aberdeen (Other); Monash University (Other)
Responsible Party: Sponsor
Other Study IDs: 16IC3652
Record Dates: First submitted 2019-08-07; First posted 2019-08-21 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2024-01

CONDITIONS: Asthma; Wheezing
Keywords: Asthma
MeSH Terms: conditions — Asthma; Respiratory Sounds

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Nasal and throat swabs, nasal epithelial cells, mRNA from nasal epithelial cells, mRNA from blood, blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- 1/Birth cohort: Prospective, longitudinal cohort of 1000 healthy infants. Recruited at birth and followed for 3 years. Samples to be collected at 5-10 days old, 1 and 3 years old. 100 participants with additional samples collected at 3 and 6 months of age. Approximately 300 participants to have samples collected at time of active wheezing and during convalescence.
- 2/mild wheezers and controls: Children under 5 years old undergoing elective general surgical procedure. Some will have mild-to-moderate wheeze while others will be non-wheezing controls
- 3/pre-school aged severe wheezers: 50 children aged 1-6 years undergoing clinically indicated bronchoscopy due to recurrent wheezing.
- 4/school aged severe asthmatics: 50 kids aged 6-16 undergoing clinically indicated bronchoscopy due to asthma.

SUMMARY:
The investigators want to know why some babies wheeze and some of these go on to develop asthma. The investigators are going to find out if babies who develop wheeze and asthma have abnormal airway lining cells (taken from the nose) when they are born and what happens to these cells as they get older.

The study will last three years. Parents will be asked to fill in a monthly health questionnaire. The tests on the babies are all in routine clinical use: a urine sample, a blood test from a heel or finger prick, swabs from the nose and throat to look at the microbiome, and a brushing of cells from the inside of the nose. These tests will be performed at 5-10 days old, and at one and three years. Parents will be asked to fill in online monthly health questionnaire. Some babies will have the swabs repeated at 3 and 6 months, and those who wheeze in the first 3 years of life, samples during the illness and after recovery.

DETAILED DESCRIPTION:
The cells that line the airways act as a barrier to infections and proteins that cause allergy, and also release a host of signalling molecules. It known that these airway cells in children with established asthma react abnormally to viruses, but not known if this is cause or consequence of asthma. Also, little is known about how the immune system develops in new born babies and how it responds to the bacteria which they meet.

This research arises from a £4.64 million Wellcome Trust strategic award. The importance of the underlying question was established with by the investigators, and the grant was developed by the collaborators at an all-day meeting followed by further telephone conferences. The Wellcome Trust also guided the development of the grant, it was peer-reviewed, it was interviewed after answering a series of questions from the referees, and subsequent to the interview, a further set of questions were answered before the Award letter was issued.

The overarching research hypothesis is that babies who develop asthma have abnormal epithelial function at birth, which further deviates from normal during the first 3 years of life. The vision is to understand what initiates asthma; facilitate development of biomarkers predicting progression of preschool wheeze to asthma; and eventually, outwith this study (in which there is no therapeutic intervention), design randomised controlled trials targeted at high risk children. The ultimate goal is preventing asthma initiation and improving lifelong lung health.

Asthma is predominantly a childhood onset disease affecting over 300 million people worldwide, and over a million children in the United Kingdom. At birth, babies who subsequently wheeze have airflow obstruction and altered immune responses. Babies who will develop asthma have airflow obstruction at birth, which worsens to age six. Thereafter, all birth cohorts have shown that lung function tracks, one of the longest (Melbourne) going on into the sixth decade of life. The first six years of life are therefore critical in determining adult lung function. Mouse data suggest that airway epithelial function is abnormal but translational evidence is lacking. Genetic and environmental factors are important in evolution of wheeze. Viral infection is a major cause of acute wheeze, but bacteria are at least as important, and early bacterial colonisation is associated with abnormal mucosal immunology. An abnormal airway microbiome skews systemic immunity to an allergic phenotype. The airway is no mere passive barrier, but also secretes innate cytokines, e.g. IL-33, which are implicated in early wheeze. Aeroallergen sensitization in the first 4 years of life, but not thereafter, is strongly predictive of subsequent asthma. Taken together, this suggests that understanding developmental changes in epithelial functions, and interactions with genes, immunity and pathogens, are crucial if progression to asthma is to be halted. The first 4 years of life represent a unique window during which adverse effects have irreversible consequences. However, understanding of the developing immune system and underlying epithelial-immune interactions during this critical period is very superficial, and it is this which the present application addresses. A significant limitation of all birth cohorts to date is the absence of airway epithelial samples to determine the mechanisms that underlie the development of early airflow obstruction and identify molecular targets for disease prevention. This project will be the first to investigate the three way interactions between airway epithelial cell function, immune responses and airway microbiota in the first four years of life to elicit the mechanisms underlying the development of preschool wheeze and its progression to asthma. The vision is to understand what initiates asthma; facilitate development of biomarkers predicting progression of pre-school wheeze to asthma; and ultimately, design interventions targeted only at high risk children, evaluated in randomised controlled trials outwith this grant. The ultimate goal is preventing asthma initiation and improvement of lifelong lung health.

Key research questions are:

1. How does epithelial function evolve from birth to 3 years in children who develop asthma, and how does the epithelium interact with the evolving immune system and airway microbiome?
2. What are the mechanisms whereby pathogens and aeroallergens modulate epithelial-immune interactions, skewing airway responses towards asthma rather than resolution?
3. Can these pathways be used to identify biomarkers of asthma development, enabling future preventive strategies?

The aims are:

1. To establish uniform clinical phenotyping and protocols for longitudinal and prospective sample acquisition
2. To utilise bioinformatics and systems biology to identify phenotypic clusters
3. To utilise an integrated clinical/basic science (systems based) approach to investigate molecular interactions between respiratory epithelium, genetics, infections, and the developing immune system and airway microbiome.

Specific objectives are:

1. Recruit newborn babies with detailed antenatal history, and obtain nasal epithelial cells at one week of age, and follow them longitudinally for three years with serial sampling, retrospectively phenotyping them depending on whether they develop wheeze or not.
2. Compare the evolving changes in immune and epithelial function in this group with the pathobiology of established mild and severe wheezers.
3. Use these samples to understand the normal and abnormal developmental interactions between the airway epithelium, the host immune system and the airway microbiome.
4. Utilize the rich longitudinal data on childhood wheezing, relevant biomarkers and genetics assembled through the birth cohorts to model the biological complexity of preschool wheezing and generate hypotheses that can be tested in vitro in age- appropriate epithelial cell cultures

ELIGIBILITY:
Inclusion Criteria:

* expectant mother or infant aged 0-10 days
* children with recurrent wheezing and other clinical atopy
* children with recurrent wheezing and no obvious wheezing triggered by aeroallergens and no clinical evidence of other atopy.
* children with no history of wheezing but with at least one clinically apparent atopic disorder
* children with no history of wheezing and with no clinical evidence of other atopic disorder
* all children will be undergoing an elective surgical procedure
* all children will have been born at term (37-42 weeks gestation)
* the anaesthetist will have deemed the child fit for elective surgery, free from a recent respiratory tract infection, stable and suitable for the research study samples to be taken.
* in the case of blind non-bronchoscopic sample suitable for endotracheal intubation or for a fibre-optic bronchoscopy if this is the chosen method of sampling

Exclusion Criteria:

* pre-term infants (<37 weeks gestation)
* twins or other multiples
* maternal group B streptococcus on high vaginal swab in the present pregnancy
* need for CPAP or ventilatory support in the neonatal period
* infants with major concurrent health problems, e.g. congenital heart disease, cystic fibrosis, those requiring special feeding regimens on account of prematurity or illness
* infants who will not be available to assess acutely if they develop wheeze
* infants who are likely to move away from the study centre before 3 years of age
* children with a recent respiratory tract illness (should have recovered > 2 weeks)
* children with other major respiratory illnesses such as and including Cystic Fibrosis, Chronic Neonatal Lung Disease, pulmonary aspiration syndromes.
* children with evidence of a systemic inflammatory or infective condition
* children with a history of previous pituitary or ethmoid surgery

Ages: 5 Days to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Singleton neonates with the developing wheeze in the before their third birthday and young children (≤5 years) with a history of mild to moderate wheezing, and those without previous wheezing.
Sampling Method: Probability Sample
Enrollment: 1300 (Estimated)
Dates: Start 2017-02-20 (Actual); Primary Completion 2024-09-18 (Estimated); Study Completion 2024-09-18 (Estimated)

PRIMARY OUTCOMES:
Changes on airway epithelium cells assessed by cell biology tools | 3 years
  To detect the airway epithelium cells differences between onset of wheeze, wheezers and non-wheezers with swabs from the nose

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Bush, MD, Principal Investigator — Imperial College London
Locations (1):
- Royal Brompton and Harefield NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No